CLINICAL TRIAL: NCT07346664
Title: Northern Jiangsu People's Hospital Affiliated to Yangzhou University
Brief Title: Medication Adherence and Lipid Management in Patients With Coronary Heart Disease After Percutaneous Coronary Intervention: Application of the Transitional Care Model
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Qing Wang (Other)
Responsible Party: Sponsor-Investigator, Qing Wang, Northern Jiangsu People's Hospital Affiliated to Yangzhou University, Northern Jiangsu People's Hospital
Organization: Northern Jiangsu People's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: No. 20240410
Record Dates: First submitted 2026-01-08; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2022-04

CONDITIONS: Transitional Care Model; Coronary Heart Disease; Medication Adherence; Self-efficacy; Lipid Profile
MeSH Terms: conditions — Coronary Disease; Medication Adherence

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- routine nursing care group (Other): Patients assigned to the control group underwent routine nursing care based on the standardized medical treatment, including admission health education (PCI postoperative risk management and medication instructions), psychological counseling, dietary and exercise guidance, individualized rehabilitation planning, and discharge instructions. After discharge, patients attended routine outpatient follow-up visits, including laboratory testing of blood lipids, blood pressure, and blood glucose, without structured follow-up or WeChat-based education. Routine outpatient education and guidance were provided only.
  Interventions: Other: routine nursing care group
- TCM intervention group (Other): Patients in the observation group received a 3-month TCM intervention delivered by specially trained nurses, in addition to routine nursing care.
  Interventions: Other: TCM intervention group

INTERVENTIONS:
Other: routine nursing care group — Patients assigned to the control group underwent routine nursing care based on the standardized medical treatment, including admission health education (PCI postoperative risk management and medication instructions), psychological counseling, dietary and exercise guidance, individualized rehabilitation planning, and discharge instructions. After discharge, patients attended routine outpatient follow-up visits, including laboratory testing of blood lipids, blood pressure, and blood glucose, without structured follow-up or WeChat-based education. Routine outpatient education and guidance were provided only.
  Arms: routine nursing care group
Other: TCM intervention group — Patients in the observation group received a 3-month TCM intervention delivered by specially trained nurses, in addition to routine nursing care.
  Arms: TCM intervention group

SUMMARY:
Patients with coronary heart disease (CHD) require long-term medication and lifestyle modification following percutaneous coronary intervention (PCI). However, they often face challenges such as poor medication adherence and inadequate self-management. This study aims to evaluate the effects of the transitional care model (TCM) on CHD patients after PCI, regarding medication adherence, self-efficacy, and lipid levels.

DETAILED DESCRIPTION:
TCM improved medication adherence, self-efficacy, and lipid profiles in CHD patients after PCI, while enhancing overall patient satisfaction. Compared with routine nursing care, TCM yielded superior clinical benefits and is recommended for broader application in the post-PCI management of CHD patients.

ELIGIBILITY:
Inclusion Criteria:

* patients clinically diagnosed with CHD according to established diagnostic criteria
* patients who met the World Health Organization (WHO) indications for PCI
* complete clinical data available

Exclusion Criteria:

* Patients with cognitive impairment
* Patients with incomplete follow-up data.
* Patients with comorbid malignancy
* Patients with severe hepatic
* Patients with renal insufficiency

Ages: 47 Years to 58 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 108 (Actual)
Dates: Start 2022-07-11 (Actual); Primary Completion 2024-05-09 (Actual); Study Completion 2024-05-26 (Actual)

PRIMARY OUTCOMES:
Medication Adherence | Baseline (before discharge) and 3 months after discharge
  Medication adherence will be assessed using the Medication Adherence Report Scale-5 (MARS-5). The scale consists of 5 items that evaluate nonadherent behaviors (e.g., forgetting to take medications, altering dosages). Each item is scored on a 5-point Likert scale (1="always" to 5="never"), with total scores ranging from 5 to 25. A higher total score indicates better medication adherence.

SECONDARY OUTCOMES:
Self-efficacy | Baseline (before discharge) and 3 months after discharge
  Self-efficacy will be assessed using the General Self-Efficacy Scale (GSS). The GSS is a validated 16-item instrument, with each item scored from 0 to 4. Higher total scores reflect greater self-efficacy in managing health and adhering to treatment recommendations.
Lipid Profile | Baseline (before discharge) and 3 months after discharge.
  Fasting serum levels of total cholesterol (TC), triglycerides (TG), high-density lipoprotein cholesterol (HDL-C), and low-density lipoprotein cholesterol (LDL-C) will be measured using an automated biochemical analyzer. All measurements will be performed in mmol/L.

CONTACTS AND LOCATIONS:
Locations (1):
- Northern Jiangsu People's Hospital Affiliated to Yangzhou University, Yangzhou, Jiangsu, China